CLINICAL TRIAL: NCT03089996
Title: Piezocision, Corticotomy and Micro-ostoeperforations to Accelerate Orthodontic Tooth Movement
Brief Title: Evaluation of Clinical Approaches to Accelerate Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontifícia Universidade Católica de Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Rodrigo Villamarim Soares, Clinical Professor, Pontifícia Universidade Católica de Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Accelerate Tooth Movement
Record Dates: First submitted 2017-01-31; First posted 2017-03-24 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Orthodontic Tooth Movement
Keywords: piezocision; corticotomy; Gingival Crevicular Fluid; Micro-osteperforations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Piezocision (Experimental): Piezocision-assisted canine retraction x Control (split mouth design)
  Interventions: Procedure: Piezocision; Device: Control Side
- Corticotomy (Experimental): Corticotomy-assisted canine retraction x Control (split mouth design)
  Interventions: Procedure: Corticotomy; Device: Control Side
- Piezocision x Corticotomy (Experimental): Piezocision-assisted retraction x Corticotomy-assisted retraction (split mouth design)
  Interventions: Procedure: Piezocision; Procedure: Corticotomy
- Micro-osteoperforations (Experimental): Micro-osteoperforations-assisted upper incisors retraction
  Interventions: Procedure: Micro-osteoperforations
- Control (No Intervention): Upper incisors retraction not associated with any clinical intervention to accelerate tooth movement

INTERVENTIONS:
Procedure: Piezocision — The first maxillary premolars will be extracted with orthodontic purpose. After 3 months of extraction, the orthodontic alignment and dental leveling will be obtained and a 0.016x0.022 stainless steel wire will be placed, as well as orthodontic mini-implants (Morelli®, Sorocaba, SP, Brazil). The retraction of the canines will begin using closed nickel-titanium spring (120g). The piezocision surgery will be performed only in one side of the mouth. Three vertical piezo-incisions will be performed near the edentulous region and mesially to the canine root, in the vestibular alveolar cortical bone with the Ultrasonic instrument (BS1 insert Piezotome ™, Satelec Group Acteon Merignac, France) in depth of 3 mm. The intraoral digital scans will be performed with 7 and 14 days after the start of retraction, and then 14 in 14 days to a maximum period of 6 months. The patients will be advised to take analgesics (paracetamol or dipyrone) only if necessary.
  Arms: Piezocision; Piezocision x Corticotomy
Procedure: Corticotomy — The first maxillary premolars will be extracted with orthodontic purpose. After 3 months of extraction, the orthodontic alignment and dental leveling will be obtained and a 0.016x0.022 stainless steel wire will be placed, as well as orthodontic mini-implants (Morelli, Sorocaba, SP, Brazil).The retraction of the canines will begin using closed nickel-titanium spring (120g).The corticotomy surgery will be performed at the day of begining of canine retraction only in one side of the mouth.A mucoperiosteal flap will be raised from the extraction region to the mesial of the canine.Perforations will be performed using a number 2 spherical drill bit in low speed handpiece under irrigation, only in the cortical none depth.The intraoral digital scans will be performed with 7 and 14 days after the start of retraction, and then 14 in 14 days to a maximum period of 6 months.The patients will be advised to take analgesics (paracetamol or dipyrone) only if necessary.
  Arms: Corticotomy; Piezocision x Corticotomy
Device: Control Side — The first maxillary premolars will be extracted with orthodontic purpose. Fixed orthodontic appliance will be bonded (0.022x0.025 slot with MBT prescription in incisors and Standart in the other teeth) with a power arm welded in the bracks upper canines brackets. After 3 months of extraction, the alignment and dental leveling will be obtained and a 0.016x0.022 stainless steel wire will be placed, as well as orthodontic mini-implants (Morelli®, Sorocaba, SP, Brazil) between the roots of the second premolars and molars. At that time an intra-oral digital scan will be performed. The retraction of the canines will begin using closed nickel-titanium spring (120g of force) from the power arm to the mini-implant. No surgery will be done at this side. The intraoral digital scans will be performed with 7 and 14 days after the start of retraction, and then 14 in 14 days to a maximum period of 6 months.
  Arms: Corticotomy; Piezocision
Procedure: Micro-osteoperforations — All micro-osteoperforations will be performed only once time in the experimental group on the same day of the installation of the upper incisors' retraction mechanics. Perforations will be performed with an individualized surgical guide and a 1.6 mm diameter stainless steel surgical drill perpendicular to the alveolar bone, 3 mm deep on the buccal surface, and 5 mm, on the palate. The depth of the perforations will be controlled and standardized by a cursor developed and patented by the research group. Two micro-osteoperforations will be aligned vertically distally from each upper incisor. Due to the proximity of the roots in the cervical third, only the most apical perforation will be performed between the two central incisors. The first perforation will be performed 6 mm away from the gingival margin, and the second, 5 mm from the first, in the vertical direction.
  Other Names: MOP
  Arms: Micro-osteoperforations

SUMMARY:
This study will compare the techniques of piezocision and alveolar corticotomies in accelerating orthodontic retraction movement of canines. In a second phase, this clinical trial will evaluate the effectiveness of micro-osteoperforations in accelerating the retraction of maxillary incisors.

DETAILED DESCRIPTION:
The first phase will consist of a split-mouth study in patients who require the extraction of the first premolars to correct malocclusion. The canine will be retracted using corticotomy and piezocision surgical techniques, as well as without any intervention, being this the control side. In addition, it will be evaluated the inflammatory biomarkers present in the gingival crevicular sulcus during the dental movement, as well as data related to pain and discomfort. The second phase will evaluate the effects of micro-osteoperforations in the retraction of maxillary incisors. The following parameters will be evaluated in the upper arch: anteroposterior incisors and first molars displacement, space closure, inclination and length of central incisors.

ELIGIBILITY:
Inclusion Criteria:

* Patient with orthodontic need for bilateral upper first premolar extraction.
* Adequate dento-oral health
* ASA I and ASA II
* Compliance with clinic visits every 2 weeks

Exclusion Criteria:

* History of periodontal disease
* Smokers
* Altered bone metabolism (e.g., due to anti-resorptive drug, steroid or immunosuppressant use)
* Pregnancy
* Presence of cleft or any syndrome

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Orthodontic Canine Retraction Rate | Up to 6 months
  The main objective is to evaluate and compare the canine retraction velocity in the different groups. Digital intra-oral scans will be performed (3Shape A / S®, Kopenhagen, Denmark) as registration method, every 14 days, up to 6 months.
Anteroposterior displacement of the upper incisors | Up to 4 months
  The anteroposterior displacement of the upper incisors was assessed on superimposed digital models through the distance of points on the incisal edge and palatal cervical margin of these teeth to a coronal reference plan created on the initial CBCT scan.
Space closure | Up to 4 months
  The space closure was assessed by the distance between the most menial point of the medial surface of the canine to the most distal point of the distal surface of the lateral incisor.

SECONDARY OUTCOMES:
Duration of the effect of the surgical procedures | Up to 6 months
  The retraction of the canine will be accompanied by up to 6 months after surgery to verify the duration of its effect, if it occurs.
Evaluation of biomarkers | Up to 6 months
  To evaluate the expression of the inflammatory biomarkers present in the gingival crevicular sulcus of the canines to be retracted. At T0, immediately before retraction, and 15 in 15 days.
Patient Pain and discomfort | Up to 6 months
  VAS questionnaire will be used after the surgical procedures, as well after TADs placement, separator placement and premolar extraction. Always 7 days after each procedure.
First molars anchorage loss | Up to 4 months
  The first molars anchorage loss was assessed on superimposed digital models through the distance of a point on the mesiobuccal cuspid to a coronal reference plan created on the initial CBCT scan.
Changes of the inclination of the central incisors | Up to 4 months
  The initial and final CBCT were superimposed by the "voxel-based method" in the Dolphin Imaging software (Chatsworth, CA, USA), using the cranial base as reference. The inclination of the central incisors was then assessed by means of the angle formed by the long axis of each central incisor in the initial and final CBCT.
Changes of the length of the central incisors | Up to 4 months
  The initial and final length of the central incisors were measured by creating a 2D line, passing through the lowest point of the incisal edge and the highest point of the root apex. To perform these measurements, a sagittal cut was used in which the longest length of these teeth was seen.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo V Soares, Phd, Study Director — Pontifícia Universidade Católica de Minas Gerais
Locations (1):
- Pontifícia Universidade Católica de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Derived] Mordente CM, Dores LS, Oliveira DD, Palomo JM, Souki BQ, Soares RV. Third Palatal Rugae as Stable Landmarks for Intraoral Models' Superimposition in Extraction Cases: A Retrospective Cohort Study. Orthod Craniofac Res. 2025 Dec 25. doi: 10.1111/ocr.70078. Online ahead of print. PMID 41445469
- [Derived] Mordente CM, Oliveira DD, Palomo JM, Cardoso PA, Assis MAL, Zenobio EG, Souki BQ, Soares RV. The effect of micro-osteoperforations on the rate of maxillary incisors' retraction in orthodontic space closure: a randomized controlled clinical trial. Prog Orthod. 2024 Feb 12;25(1):6. doi: 10.1186/s40510-023-00505-z. PMID 38342823
- [Derived] Fernandes LSDMCP, Figueiredo DSF, Oliveira DD, Houara RG, Rody WJ Jr, Gribel BF, Soares RV. The effects of corticotomy and piezocision in orthodontic canine retraction: a randomized controlled clinical trial. Prog Orthod. 2021 Oct 4;22(1):37. doi: 10.1186/s40510-021-00367-3. PMID 34604918